CLINICAL TRIAL: NCT05135585
Title: Evaluation of the Post-vaccination Immune Response to COVID-19 in the New Caledonian Population
Acronym: COVCAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Centre Hospitalier Spécialisé de Nouvelle-Calédonie (Unknown); Direction de l'Action Sanitaire et Sociale (Other Government); Centre Hospitalier Territorial de Nouvelle-Calédonie (Other); Agence sanitaire et sociale de la Nouvelle Calédonie (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-059; 2021-A01949-32 (Other: ID-RCB)
Record Dates: First submitted 2021-11-23; First posted 2021-11-26 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2021-10

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease
Keywords: Immune Response; Vaccination; Pacific; Population of New Caledonia
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults vaccinated with a complete COVID-19 vaccine regimen (Other): Adults of Melanesian, Polynesian, European, and other communities vaccinated with a complete COVID-19 vaccine regimen, residing in New Caledonia.
  Interventions: Other: Blood sample collection; Other: Questionnaires

INTERVENTIONS:
Other: Blood sample collection — Blood sample collection at 1 month and 6 months after vaccination
Other: Questionnaires — data collection (health data, vaccination data, etc.)

SUMMARY:
The COVID-19 pandemic caused by SARS-CoV-2 since December 2019 has caused more than 210 million cases worldwide as of September 1, 2021. New Caledonia (NC) is an ultramarine French territory in the South Pacific so far relatively spared by this pandemic thanks to the establishment of a health lock. The vaccination campaign started locally on 20/01/2021 with the exclusive use of Pfizer's COMIRNATY mRNA vaccine. Vaccination is now offered to anyone over the age of 12. Vaccination against COVID-19 will be mandatory in New Caledonia as of October 31, 2021 for certain exposed populations and for the entire adult population as of December 31, 2021.

Clinical trials of COVID-19 vaccines, including those of mRNA vaccines, have taken care to maintain ethnic diversity within their samples. Efficacy studies have not shown a significant difference in the efficacy of Pfizer COMIRNATY vaccine in white, black American, or Hispanic populations. The response of non-European non-Asian Oceanian populations to Pfizer COMIRNATY vaccination has not been specifically studied at this time. According to the 2019 census in New Caledonia, 41.2% of the population identified themselves as Kanak (Melanesian), 24% as European, 8.3% as Wallisian-Futunian (Polynesian), 11% as mestizo, and 8% as belonging to other communities including Tahitian (Polynesian), Indonesian, Ni-Vanuatu (Melanesian), and Vietnamese communities (8). Some recent data are in favor of a significant variability of susceptibility to pathogens in Oceanian populations, stemming from a genetic inheritance from Neanderthal man and his cousin Denisova man. In a context of vaccine hesitancy, it is therefore important to ensure that the immune response of the New Caledonian population (Melanesian, Polynesian, European or other communities) to vaccination against COVID-19 is similar to that of populations studied in large clinical trials.

DETAILED DESCRIPTION:
Observational equivalence study with prospective data collection. Vaccinated subjects to be included will be identified in the vaccination centers in the Southern Province during the injection of the second dose.

Information and consent collection. Completion of a questionnaire and collection of 4 mL of blood on a dry tube at M1 and M6 months.

Testing for the presence of anti-SARS-CoV-2 antibodies by ELISA (anti-Spike and anti-Nucleoprotein).

Return of the results of the serological analyses to the participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults from Melanesian, Polynesian, European or other community origin
* Adults vaccinated with 2 doses of Pfizer COMIRNATY vaccine, administered between 3 and 12 weeks apart
* Adults planning to be present in the territory and to be available on both sampling dates (1 and 6 months)

Exclusion Criteria:

* Persons who received the second dose of vaccine more than 12 weeks after the first dose
* Persons vaccinated against COVID-19 with a vaccine other than Pfizer COMIRNATY
* Women who report being pregnant or breastfeeding (where the immune response may be altered)
* Immunocompromised persons (immunosuppressive treatment, immunomodulator, HIV positive, splenectomy, long term corticosteroid therapy, autoimmune diseases such as rheumatoid arthritis, lupus, spondyloarthritis, etc.)
* People who are not intellectually capable of answering the questionnaire
* Persons under guardianship, curatorship or any other legal incapacity
* Persons with documented Covid-19 infection (known positive SARS-CoV-2 serology prior to inclusion, positive PCR or antigen test)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-09-17 (Actual); Study Completion 2022-09-17 (Actual)

PRIMARY OUTCOMES:
Measurement by ELISA tests of the presence of antibodies at 1 month after the second dose of Pfizer COMIRNATY vaccine in the New Caledonian population | 6 months
  To assess in a standardized manner the humoral immune response to COVID-19 vaccination at 1 month after the second dose in vaccinated individuals of Polynesian, Melanesian, European and other communities in New Caledonia

SECONDARY OUTCOMES:
Measurement by ELISA of the presence of antibodies at 6 months after the second dose of Pfizer COMIRNATY vaccine in the New Caledonian population | 1 year
  To evaluate and compare in a standardized manner the humoral immune response to COVID-19 vaccinationat 6 months after the second dose of Pfizer COMIRNATY vaccine in vaccinated individuals of Polynesian, Melanesian, European and other communities in New Caledonia
Serum neutralization analysis of the neutralizing capacity against different circulating SARS-CoV-2 variants of antibodies secreted at 1 and 6 months after the second dose of Pfizer COMIRNATY vaccine in the New Caledonian population | 1 year
  To study the functionality (neutralizing capacity) of antibodies secreted in response to COVID-19 vaccination by individuals of Melanesian, Polynesian, European and other community origin at 1 month and 6 months after the second dose of Pfizer COMIRNATY vaccine
Post-hoc analysis of anti-Spike and anti-Nucleoprotein ELISA results at 1 month by age stratification (group over 70 years and control group 20-59 years) | 1 year
  To evaluate and compare in a standardized way the humoral immune response to the COVID-19 vaccination at 1 month after the second dose of Pfizer COMIRNATY vaccine in subjects aged over 70 years and a control group in the New Caledonian population

CONTACTS AND LOCATIONS:
Overall Officials: Myrielle Dupont-Rouzeyrol, PhD, Study Director — Institut Pasteur de Nouvelle-Calédonie; Valérie Albert-Dunais, MD, Principal Investigator — Centre Hospitalier Spécialisé de Nouvelle-Calédonie
Locations (3):
- New Caledonia (3):
  - Centre Hospitalier Territorial de Nouvelle-Calédonie, Dumbéa Sur Mer
  - Centre hospitalier spécialisé de Nouvelle-Calédonie, Noumea
  - Vaccination centers, Province Sud

REFERENCES:
- [Derived] Inizan C, Courtot A, Sturmach C, Griffon AF, Biron A, Bruel T, Enouf V, Demaneuf T, Munier S, Schwartz O, Gourinat AC, Medevielle G, Jouan M, van der Werf S, Madec Y, Albert-Dunais V, Dupont-Rouzeyrol M. Levels and functionality of Pacific Islanders' hybrid humoral immune response to BNT162b2 vaccination and delta/omicron infection: A cohort study in New Caledonia. PLoS Med. 2024 Sep 26;21(9):e1004397. doi: 10.1371/journal.pmed.1004397. eCollection 2024 Sep. PMID 39325828